CLINICAL TRIAL: NCT06243055
Title: Reliability and Validity of the Turkish Version of the Laval Quality of Life Questionnaire for Obesity
Brief Title: Reliability and Validity of the Turkish Version of the Laval
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, İzmir Bayraklı District Health Directorate, Ege University
Other Study IDs: 6617-GOA
Record Dates: First submitted 2024-01-16; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Quality of Life
Keywords: obesity; quality of life; validity and reliability
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnare — laval questionnare
Other: questionnare — Obese-Specific Quality of Life
Other: questionnare — SF-12 Quality of Life scale

SUMMARY:
The study is a Turkish validity and reliability study of the Laval questionnaire.

DETAILED DESCRIPTION:
the study was planned as a student's master thesis. the whole study was carried out by us. all evaluations were completed. all analyses were completed. It is an observational study. It is a survey study.The study data were entered retrospectively.

Research İzmir Bayraklı District Health Directorate No. 1 Healthy Life Centre (1 October 2021 - 15 November 2021) and Gaziemir Municipality (15 November 2021 - 15 March 2022) was conducted. Dokuz Eylül University Ethics Committee accepted the study on 22.12.2021 with the decision number 2021/38-08. People with Body Mass Index ≥ 30 kg/m2 and who met the inclusion/exclusion criteria were included in the study. In addition to the Laval Questionnaire, the SF-12 general health quality of life questionnaire and the Obese-Specific Quality of Life Scale were used. For the adaptation of the Turkish version of the questionnaire, first, language validity was ensured by back translation method.

ELIGIBILITY:
Inclusion Criteria:

* volunteering, being literate
* age ≥ 18 and age ≤ 75
* body mass index (BMI) ≥ 30 kg/m2
* ability to follow instructions to fill out questionnaires.

Exclusion Criteria:

* affected by psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: body mass index (BMI) ≥ 30 kg/m2
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
the Kaiser-Meyer-Olkin (KMO) test | 1 year
  to check the suitability of the sample number for analysis

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziemir Municipality, Izmir, Gaziemir
  - İzmir Bayraklı District Health Directorate No. 1 Healthy Life Centre, Bayraklı, İ̇zmi̇r

IPD SHARING:
Plan to Share IPD: Yes
In addition to the Laval Questionnaire, the SF-12 general health quality of life questionnaire and the Obese-Specific Quality of Life Scale were used.
Supporting Information: Study Protocol
Time Frame: Research İzmir Bayraklı District Health Directorate No. 1 Healthy Life Centre (1 October 2021 - 15 November 2021) and Gaziemir Municipality (15 November 2021 - 15 March 2022) was conducted